CLINICAL TRIAL: NCT05959109
Title: A Phase 1, Single-Dose Study to Assess the Relative Bioavailability and Tolerability of Subcutaneous Peresolimab Test Formulations in Healthy Participants
Brief Title: A Relative Bioavailability Study of Peresolimab (LY3462817) Formulations in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 18608; J1A-MC-KDAI (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-07-17; First posted 2023-07-25 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Peresolimab (Test 1) (Experimental): Peresolimab administered subcutaneously (SC).
  Interventions: Drug: Peresolimab
- Peresolimab (Test 2) (Experimental): Peresolimab administered SC.
  Interventions: Drug: Peresolimab
- Peresolimab (Test 3) (Experimental): Peresolimab administered SC.
  Interventions: Drug: Peresolimab
- Peresolimab (Reference) (Experimental): Peresolimab administered SC.
  Interventions: Drug: Peresolimab

INTERVENTIONS:
Drug: Peresolimab — Administered SC
  Other Names: LY3462817

SUMMARY:
The main purpose of this study is to look at the amount of the study drug, peresolimab, that gets into the blood stream and how long it takes the body to get rid of it when given under the skin using test formulations versus reference formulation in healthy participants. The study will also evaluate the safety and tolerability of peresolimab and information about any side effects experienced will be collected. For each participant, the total duration of the study will be approximately up to 17 weeks, including screening.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants who are overtly healthy as determined by medical history, physical examination, and other screening procedures
* A minimum body weight of 45 kilograms and body mass index (BMI) between 18.0 and 32.0 kilograms per meter squared (kg/m²), inclusive, at screening
* Have blood pressure, pulse rate, blood and urine laboratory test results that are acceptable for the study
* Males who agree to use highly effective/effective methods of contraception and women not of childbearing potential

Exclusion Criteria:

* Have significant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs, of constituting a risk when taking the study intervention, or of interfering with the interpretation of data
* Have a history of allergy to monoclonal antibody therapy or to the excipients in the drug formulation, or have clinically significant intolerance to topical corticosteroids, or a history of severe posttreatment hypersensitivity reactions (including, but not limited to, erythema multiforme major, linear IgA dermatosis, toxic epidermal necrolysis, or exfoliative dermatitis).
* Have a diagnosis or history of malignant disease within 5 years prior to screening, with the following exceptions:

  1. basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years
  2. cervical carcinoma in situ, with no evidence of recurrence within the 5 years prior to screening.
* Are immunocompromised.
* Have known hypogammaglobulinemia
* Have a current or recent acute, active infection. For at least 30 days before screening and up to the baseline visit, participants must have no symptoms or signs of confirmed or suspected infection and must have completed any appropriate anti-infective treatment.
* Have had any of the following types of infection within 3 months prior to the screening visit or develops any of these infections before the baseline visit:

  1. serious (requiring hospitalization, or IV or equivalent oral antibiotic treatment, or both)
  2. opportunistic (as defined in Winthrop et al. 2015)
  3. chronic (duration of symptoms, signs, and/or treatment of 6 weeks or longer)
  4. recurring (including, but not limited to, herpes simplex, herpes zoster, recurring cellulitis, chronic osteomyelitis).
* Have active TB.
* Have or have had latent tuberculosis infection that has not been treated with a complete course of appropriate therapy as defined by the World Health Organization and the United States Centers for Disease Control and Prevention, unless such treatment is underway.
* Have a current infection with HBV (that is, positive for hepatitis B surface antigen and/or polymerase chain reaction positive for HBV DNA).
* Have a current infection with HCV (that is, positive for HCV RNA).
* Have HIV infection.
* Have received treatment with biologic agents (such as monoclonal antibodies, including marketed drugs) within 3 months or 5 half-lives (whichever is longer) prior to dosing.
* Have received any live vaccine (that is, live attenuated) within less than 4 weeks before screening or intend to receive a live vaccine during the study, or within 5 half-lives (8 weeks) after receiving the last dose of study intervention, whichever is longer. Note: The following are not considered live vaccines: RNA vaccines, vaccines with inactive viral elements, and/or nonreplicating viral vector vaccines.
* Have received a bacille Calmette-Guerin vaccination or treatment within less than 4 weeks before screening or intend to receive bacille Calmette-Guerin vaccination or treatment during the study, or within 5 half-lives (8 weeks) after receiving the last dose of study intervention, whichever is longer.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2023-07-21 (Actual); Primary Completion 2024-01-11 (Actual); Study Completion 2024-01-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Maximum Concentration (Cmax) of Peresolimab | Predose up to 85 days postdose
  PK: Cmax of Peresolimab
PK: Area Under the Plasma Concentration Versus Time Curve from Zero to T, Last Time Point (AUC[0-tlast]) of Peresolimab | Predose up to 85 days postdose
  PK: AUC[0-tlast] of Peresolimab
PK: Area Under the Plasma Concentration Versus Time Curve From Zero to Infinity (AUC[0-∞]) of Peresolimab | Predose up to 85 days postdose
  PK: AUC(0-∞) of Peresolimab

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- LabCorp CRU, Inc., Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No